CLINICAL TRIAL: NCT03659422
Title: Dietary Approach to Improving QoL in ALS
Brief Title: Dietary Approach to Improving Quality of Life in Amyotrophic Lateral Sclerosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: not funded
Sponsor: Terry L. Wahls (Other)
Collaborators: Muscular Dystrophy Association (Other)
Responsible Party: Sponsor-Investigator, Terry L. Wahls, Clinical Professor of Medicine, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201802746
Record Dates: First submitted 2018-04-12; First posted 2018-09-06 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Diet Modification; Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Other): Modified Paleolithic diet and vitamin/ supplement program was part of previous approaches to managing ALS related symptoms over an 18 month period. This is a safety study. We will be assessing if patients can implement the proposed modified Paleolithic diet (Wahls Elimination), if lean muscle mass is maintained on the study diet, and what changes occur in the ALS functional symptoms and quality of life.
  Interventions: Other: Modified Paleolithic diet

INTERVENTIONS:
Other: Modified Paleolithic diet — The diet eliminates legumes, grains and nightshades (as opposed to the Paleolithic diet) and is higher in vegetable and fruit intake and in omega-3 fatty rich foods.

SUMMARY:
We have had reports of an individual who utilized a modified Paleolithic diet and vitamin/ supplement program as part of his approach to managing ALS related symptoms. This individual has experienced stability in his ALS functional rating score and stable to improving strength over an 18 month period. There are also anecdotal reports of ALS patients who have utilized a dietary approach based on a Paleolithic eating plan of improved function. This is a safety study. We will be assessing if patients can implement the proposed modified Paleolithic diet (Wahls Elimination), if lean muscle mass is maintained on the study diet, and what changes occur in the ALS functional symptoms and quality of life.

DETAILED DESCRIPTION:
Study visits: 3 total over 12 weeks. Screening prior to enrollment will include consent to complete three 24-hour dietary recalls prior to the first study visit.

Visit 0. Subject will be seen in the University of Iowa Hospitals and Clinics (UIHC) Neurology Clinic, prevention intervention center or clinical research unit to review the consent, answer questions and sign the consent.

Subjects will provide phone numbers and best times for the dietitian to call for the dietary recall interviews and will be given a 2-dimensional food portion booklet to assist with reporting amount of food eaten.

Letters and a copy of the study consent will be sent to eligible ALS patients from the UIHC ALS clinic with follow up calls as previously descried.

Questions will be answered, the consent will be reviewed. If the patient wants to participate in the study, a Visit 1 will be scheduled and permission to complete the 24 hour dietary recalls will be obtained.

Height and weight will be documented from the participant clinic visits (neurology and primary care if needed) to obtain at least 2 weights and a height obtained in a clinic setting in the prior 6 months to calculate a slope of projected weight loss per month and a projected weight loss and muscle mass loss that may be observed at visit 2.

Visit 1. Subjects will be asked to fast for 12 hours prior to visit. Urine specific gravity will be obtained. The target is 1.004 to 1.028. If the urine is too dilute, the patient is to stop drinking and the other tests will be obtained and urine specific gravity will be repeated. The urine specific gravity that is noted that is within the range -- will be the target specific gravity for future BIS tests (ideally within .005). Patients are asked to report with the same level of hydration for future tests. Resting energy expenditure, forced vitality capacity and hand grip test will be completed. Fasting blood specimens and vital signs will be obtained. Subjects will be provided with a snack (or asked to bring a snack). Questionnaires will be completed. Subjects will be educated how the subject's personal family history (genetic vulnerability) may have interacted with the patient's unique DNA and lifetime of diet, lifestyle choices and environmental exposures to contributed to the participants' current health circumstances. The subject will be instructed on a stress-reducing practice on mindfulness and the subject will do a practice session of mindfulness. The participant will be taught the study diet by the intervention dietitian. A diet checklist that offers guidance to the subject in the form of prompts to eat the foods that are recommended and to avoid those that are not recommended will be provided. The subject and their adult companion will be given a study-compliant meal and will practice recording the meal in the diet checklist to facilitate the learning of the principles of the study diet and how to use the daily diet checklist. The subject and adult companion will be instructed on mindful eating.

The study visit will take approximately 5 to 6 hours. The subject will be given a 'loaner' food blending machine to use to make smoothies and soups that are compliant with the study diet. The subject will be asked to add 20 grams of bone broth protein powder and consume that in a study compliant smoothie or warm beverage each day to increase protein intake in a food or beverage item that does not require chewing (such as a smoothie or soup.

After the study visit:

Subjects will work by telephone with the study dietitian as they implement the study diet and stress reducing practice. The subject will be called 2 to 3 days after the visit by the study dietitian to review the study diet and answer questions. The dietitian will call again in one week to review the study diet with the study subject and ask how the participant is managing the diet. The dietitian will ask the participant if they are willing to continue on the study diet for the remainder of the study which is called the intervention phase of the study. If he participant is willing to continue the study diet, they will begin adding the various vitamins and supplements according to schedule in the diet checklist. If the participant does not wish to continue the study diet, the coaching calls will stop. Even if the participant resumes their usual diet, the participant will still come in for the end of study visit 3 at 12 weeks. The participant will not come back for 12 week visit.

Visit 2: 6 weeks.

Subjects will be asked to fast for 12 hours prior to visit. The patient will be weighed. Urine specific gravity will be obtained. The target urine specific gravity for the patient future BIS tests (ideally within .005) from the first BIS will be identified. A urine sample will be obtained The urine specific gravity will be obtained and compared to the target value. If the urine is too dilute, the patient is to stop drinking and the other tests will be obtained and urine specific gravity will be repeated in 1 hour.

The changes in muscle mass between visit 1 and visit 2 will be calculated and compared to the projected muscle mass loss. If the participant has lost more muscle mass than was projected, the study dietitian will instruct the participant on strategies to increase calories and protein while following the study diet. In addition, the participant will be asked to increase the intake of bone broth protein to 40 grams per day.

This visit will take 3 hours.

Visit 3: End of Study visit at 12 weeks. Participants will return the blending machine. The target urine specific gravity for the patient future BIS tests (ideally within .005) from the first BIS will be identified. A urine sample will be obtained The urine specific gravity will be obtained and compared to the target value. If the urine is too dilute, the patient is to stop drinking and the other tests will be obtained and urine specific gravity will be repeated in 1 hour. Patients are asked to report with the same level of hydration for future tests.

Resting energy expenditure, forced vitality capacity and BIS will be completed. Fasting blood specimens and vital signs will be obtained. Subjects will be able to eat a snack. The hand grip test will be completed. Questionnaires will be completed. The study team will answer questions about the study. Three 24 hour recalls will be completed in the week before and or the week after the end of study visit.

The changes in muscle mass between visit 1 and visit 2 will be calculated and compared to the projected muscle mass loss. The participant will be informed if the muscle mass is greater than projected and will be informed of strategies to increase calorie and protein intake.

The study visit will take approximately 2 to 3 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of clinically possible, clinically probable (with or without laboratory support), or clinically definite ALS (using the revised El Escorial Criteria)
2. Ability to prepare, or have prepared for them, home-cooked meals
3. Age between 18 and 80 years
4. Followed by ALS clinic at the University of Iowa
5. Willingness to adopt the study diet

Exclusion Criteria:

1. Clinically significant liver, kidney, or heart disease
2. Taking insulin or Coumadin
3. Ventilator dependence
4. Psychiatric disorder making dietary compliance difficult (e.g. schizophrenia)
5. Unwillingness to have blood specimens collected
6. Dysphagia present
7. Greater than two years since onset of ALS symptoms

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in total body weight from baseline over 12 weeks. | 12 weeks
  body weight (kilograms)
Change in Body Mass Index from baseline over 12 weeks. | 12 weeks
  body weight (in kilograms) divided by height square (in meters)
change in fat mass (in kilograms) from baseline over 12 weeks | 12 weeks
  Bio-electrical impedance measurement of body composition
change in fat-free mass (in kilograms) from baseline over 12 weeks | 12 weeks
  Bio-electrical impedance measurement of body composition

SECONDARY OUTCOMES:
change in motor function over 12 weeks | 12 weeks
  Grip strength
change in breathing function over 12 weeks | 12 weeks
  Forced Expiratory Volume
Change in fatigue level | 12 weeks
  Fatigue Severity Scale is used. scale has 9 questions, each could range from 1 to 7. Sum responses and divide by number of items for scale score. Higher score indicates more disability.

CONTACTS AND LOCATIONS:
Overall Officials: Terry L Wahls, MD, Principal Investigator — University of Iowa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Milonas I. Amyotrophic lateral sclerosis: an introduction. J Neurol. 1998 Aug;245 Suppl 2:S1-3. doi: 10.1007/s004150050640. PMID 9747926
- [Background] Talbott EO, Malek AM, Lacomis D. The epidemiology of amyotrophic lateral sclerosis. Handb Clin Neurol. 2016;138:225-38. doi: 10.1016/B978-0-12-802973-2.00013-6. PMID 27637961
- [Background] Wang MD, Little J, Gomes J, Cashman NR, Krewski D. Identification of risk factors associated with onset and progression of amyotrophic lateral sclerosis using systematic review and meta-analysis. Neurotoxicology. 2017 Jul;61:101-130. doi: 10.1016/j.neuro.2016.06.015. Epub 2016 Jul 1. PMID 27377857
- [Background] Okamoto K, Kihira T, Kobashi G, Washio M, Sasaki S, Yokoyama T, Miyake Y, Sakamoto N, Inaba Y, Nagai M. Fruit and vegetable intake and risk of amyotrophic lateral sclerosis in Japan. Neuroepidemiology. 2009;32(4):251-6. doi: 10.1159/000201563. Epub 2009 Feb 11. PMID 19209004
- [Background] Jin Y, Oh K, Oh SI, Baek H, Kim SH, Park Y. Dietary intake of fruits and beta-carotene is negatively associated with amyotrophic lateral sclerosis risk in Koreans: a case-control study. Nutr Neurosci. 2014 Apr;17(3):104-8. doi: 10.1179/1476830513Y.0000000071. Epub 2013 Nov 26. PMID 23710627
- [Background] Fitzgerald KC, O'Reilly EJ, Falcone GJ, McCullough ML, Park Y, Kolonel LN, Ascherio A. Dietary omega-3 polyunsaturated fatty acid intake and risk for amyotrophic lateral sclerosis. JAMA Neurol. 2014 Sep;71(9):1102-10. doi: 10.1001/jamaneurol.2014.1214. PMID 25023276
- [Background] Appel SH, Smith RG, Engelhardt JI, Stefani E. Evidence for autoimmunity in amyotrophic lateral sclerosis. J Neurol Sci. 1994 Jul;124 Suppl:14-9. doi: 10.1016/0022-510x(94)90171-6. PMID 7807136
- [Background] Appel SH, Smith RG, Engelhardt JI, Stefani E. Evidence for autoimmunity in amyotrophic lateral sclerosis. J Neurol Sci. 1993 Sep;118(2):169-74. doi: 10.1016/0022-510x(93)90106-9. PMID 8229065
- [Background] Brown KJ, Jewells V, Herfarth H, Castillo M. White matter lesions suggestive of amyotrophic lateral sclerosis attributed to celiac disease. AJNR Am J Neuroradiol. 2010 May;31(5):880-1. doi: 10.3174/ajnr.A1826. Epub 2009 Nov 12. PMID 19910450
- [Background] Gadoth A, Nefussy B, Bleiberg M, Klein T, Artman I, Drory VE. Transglutaminase 6 Antibodies in the Serum of Patients With Amyotrophic Lateral Sclerosis. JAMA Neurol. 2015 Jun;72(6):676-81. doi: 10.1001/jamaneurol.2015.48. PMID 25867286
- [Background] Rao TV, Tharakan JK, Jacob PC. Systemic lupus erythematosus presenting as amyotrophic lateral sclerosis. Clin Neuropathol. 2004 May-Jun;23(3):99-101. PMID 15200286
- [Background] Maldonado ME, Williams RC Jr, Adair JC, Hart BL, Gregg L, Sibbitt WL Jr. Neuropsychiatric systemic lupus erythematosus presenting as amyotrophic lateral sclerosis. J Rheumatol. 2002 Mar;29(3):633-5. PMID 11908583
- [Background] Turner MR, Goldacre R, Ramagopalan S, Talbot K, Goldacre MJ. Autoimmune disease preceding amyotrophic lateral sclerosis: an epidemiologic study. Neurology. 2013 Oct 1;81(14):1222-5. doi: 10.1212/WNL.0b013e3182a6cc13. Epub 2013 Aug 14. PMID 23946298
- [Background] Park Y, Park J, Kim Y, Baek H, Kim SH. Association between nutritional status and disease severity using the amyotrophic lateral sclerosis (ALS) functional rating scale in ALS patients. Nutrition. 2015 Nov-Dec;31(11-12):1362-7. doi: 10.1016/j.nut.2015.05.025. Epub 2015 Jul 6. PMID 26429656
- [Background] Bouteloup C, Desport JC, Clavelou P, Guy N, Derumeaux-Burel H, Ferrier A, Couratier P. Hypermetabolism in ALS patients: an early and persistent phenomenon. J Neurol. 2009 Aug;256(8):1236-42. doi: 10.1007/s00415-009-5100-z. Epub 2009 Mar 22. PMID 19306035
- [Background] Roubeau V, Blasco H, Maillot F, Corcia P, Praline J. Nutritional assessment of amyotrophic lateral sclerosis in routine practice: value of weighing and bioelectrical impedance analysis. Muscle Nerve. 2015 Apr;51(4):479-84. doi: 10.1002/mus.24419. Epub 2015 Feb 24. PMID 25130859
- [Background] Ngo ST, Steyn FJ, McCombe PA. Body mass index and dietary intervention: implications for prognosis of amyotrophic lateral sclerosis. J Neurol Sci. 2014 May 15;340(1-2):5-12. doi: 10.1016/j.jns.2014.02.035. Epub 2014 Mar 3. PMID 24629478
- [Background] Salvioni CC, Stanich P, Almeida CS, Oliveira AS. Nutritional care in motor neurone disease/ amyotrophic lateral sclerosis. Arq Neuropsiquiatr. 2014 Feb;72(2):157-63. doi: 10.1590/0004-282X20130185. PMID 24604371
- [Background] Fitzgerald KC, O'Reilly EJ, Fondell E, Falcone GJ, McCullough ML, Park Y, Kolonel LN, Ascherio A. Intakes of vitamin C and carotenoids and risk of amyotrophic lateral sclerosis: pooled results from 5 cohort studies. Ann Neurol. 2013 Feb;73(2):236-45. doi: 10.1002/ana.23820. Epub 2013 Jan 29. PMID 23362045
- [Background] Bisht B, Darling WG, Grossmann RE, Shivapour ET, Lutgendorf SK, Snetselaar LG, Hall MJ, Zimmerman MB, Wahls TL. A multimodal intervention for patients with secondary progressive multiple sclerosis: feasibility and effect on fatigue. J Altern Complement Med. 2014 May;20(5):347-55. doi: 10.1089/acm.2013.0188. Epub 2014 Jan 29. PMID 24476345
- [Background] Lee JE, Bisht B, Hall MJ, Rubenstein LM, Louison R, Klein DT, Wahls TL. A Multimodal, Nonpharmacologic Intervention Improves Mood and Cognitive Function in People with Multiple Sclerosis. J Am Coll Nutr. 2017 Mar-Apr;36(3):150-168. doi: 10.1080/07315724.2016.1255160. Epub 2017 Apr 10. PMID 28394724
- [Background] Coyne N, Correnti D. Effectiveness of motivational interviewing to improve chronic condition self-management: what does the research show us? Home Healthc Nurse. 2014 Jan;32(1):56-63. doi: 10.1097/NHH.0000000000000001. PMID 24326477
- [Background] Vansteenkiste M, Williams GC, Resnicow K. Toward systematic integration between self-determination theory and motivational interviewing as examples of top-down and bottom-up intervention development: autonomy or volition as a fundamental theoretical principle. Int J Behav Nutr Phys Act. 2012 Mar 2;9:23. doi: 10.1186/1479-5868-9-23. PMID 22385828
- [Background] Inam S, Vucic S, Brodaty NE, Zoing MC, Kiernan MC. The 10-metre gait speed as a functional biomarker in amyotrophic lateral sclerosis. Amyotroph Lateral Scler. 2010 Dec;11(6):558-61. doi: 10.3109/17482961003792958. Epub 2010 Jun 2. PMID 20515425
- [Background] Martin JL, Hakim AD. Wrist actigraphy. Chest. 2011 Jun;139(6):1514-1527. doi: 10.1378/chest.10-1872. PMID 21652563
- [Background] Kaufmann P, Levy G, Thompson JL, Delbene ML, Battista V, Gordon PH, Rowland LP, Levin B, Mitsumoto H. The ALSFRSr predicts survival time in an ALS clinic population. Neurology. 2005 Jan 11;64(1):38-43. doi: 10.1212/01.WNL.0000148648.38313.64. PMID 15642901
- [Background] Simmons Z, Felgoise SH, Bremer BA, Walsh SM, Hufford DJ, Bromberg MB, David W, Forshew DA, Heiman-Patterson TD, Lai EC, McCluskey L. The ALSSQOL: balancing physical and nonphysical factors in assessing quality of life in ALS. Neurology. 2006 Nov 14;67(9):1659-64. doi: 10.1212/01.wnl.0000242887.79115.19. PMID 17101900
- [Background] Chio A, Gauthier A, Calvo A, Ghiglione P, Mutani R. Caregiver burden and patients' perception of being a burden in ALS. Neurology. 2005 May 24;64(10):1780-2. doi: 10.1212/01.WNL.0000162034.06268.37. PMID 15911811
- [Background] Bisht B, Darling WG, Shivapour ET, Lutgendorf SK, Snetselaar LG, Chenard CA, Wahls TL. Multimodal intervention improves fatigue and quality of life in subjects with progressive multiple sclerosis: a pilot study. Degener Neurol Neuromuscul Dis. 2015;5:19-35. doi: 10.2147/DNND.S76523. Epub 2015 Feb 27. PMID 30728736
- [Background] Irish AK, Erickson CM, Wahls TL, Snetselaar LG, Darling WG. Randomized control trial evaluation of a modified Paleolithic dietary intervention in the treatment of relapsing-remitting multiple sclerosis: a pilot study. Degener Neurol Neuromuscul Dis. 2017 Jan 4;7:1-18. doi: 10.2147/DNND.S116949. eCollection 2017. PMID 30050374